CLINICAL TRIAL: NCT02615548
Title: Investigating the Effect of Specific, Long- Term, Community-based Exercises on Walking, Balance, and Quality of Life in Adults With Parkinson Disease.
Brief Title: Exercise for Adults With Parkinson Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver Coastal Health (Other Government)
Responsible Party: Principal Investigator, Diana Krasteva, Physiotherapist, University of British Columbia
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: H15-01772
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Parkinson Disease
Keywords: exercises
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Community exercise class (Experimental): Regular community exercise class is the intervention. It is an exercise class that incorporate PWR moves( UP,ROCK,STEP,TWIST) and cardiovascular training.
  Interventions: Other: community-based exercise class
- self-directed exercise activity (Active Comparator): Self-directed exercise.
  Interventions: Other: self-directed physical activity

INTERVENTIONS:
Other: community-based exercise class — This intervention will be held in a community centre, twice per week, for 36 weeks.The participants will have an educational session regarding importance of regular exercise.The class will consist of evidence-based exercises such as: sustained, high effort exercises, resistance exercises, and endurance training.Two trainers with specific for Parkinson Disease training will lead the class.
  Arms: Community exercise class
Other: self-directed physical activity — Participants from this group will have an educational session regarding importance of regular exercises for Parkinson Disease and will be asked to stay as active as possible.Both groups will be asked to fill out physical activity diary.
  Arms: self-directed exercise activity

SUMMARY:
Physical activity is a key intervention used to reduce the healthcare costs and the negative consequences of Parkinson Disease (PD) by improving walking and balance and reducing the number of falls. However, not all exercise classes provide the same results for people with PD. Specific exercises designed to target the features of PD have shown greater outcomes than generic physical activity. The exercise principles include high-intensity (size and speed) movement, task repetition, rhythmical rocking, mental imagery, cognitive strategies, treadmill walking, and making use of internal and external cues. Collectively these PD-specific exercises can be designed to be run in exercise groups. Structured exercise groups also include social interaction that is known to improve depression and apathy, both of which are features common in people with PD.

This study will compare the effect of specific, long-term community-based exercise class on balance, walking, quality of life, and mood compare to self-directed exercise.

Investigators anticipate that participants from the community-based, long-term intervention will show better improvements in balance and walking compare to participants that are self-directing their activities.

DETAILED DESCRIPTION:
This is a mixed-method, randomized design study. Participants will be assessed using qualitative and quantitative measures before and after a nine-month intervention.Outcome measures for motor function will be described using Paired t-tests for continuous variables and McNemar's Test for categorical variables. Participants will be recruited from the LGH NROP program, North Shore physicians, and the Pacific Parkinson's Research Centre Movement Disorders Clinic, UBC. Potential participants will be approached by their treating physicians during their clinical visits. People who are interested in participating in the study will be invited to contact the NROP Registered Nurse (RN) to discuss study participation and review the inclusion and exclusion criteria. The study will recruit fifteen participants for the intensive community-based exercise group and fifteen for the self-directed exercise group.The sample size calculation was performed using G*power 3.1.9.2.Once participants provide a signed informed consent they will be randomly assigned to one of the groups by picking a number from 00 to 30 out of an envelope.

The class will consist of evidence-based exercises such as: sustained, high effort exercises, resistance exercises, and endurance training. The other participants will continue on their own. All participants will be asked to fill out a physical activity diary regarding the frequency, duration, and intensity of the activities during the nine months trial.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic PD
* Hoehn & Yahr stages 1 to 3 (17).These stages define early to mid-stage of PD.
* Adult men and/or women, age 45-80
* Willing and able to participate in 60-minute of physical activity, 3/week for 12-weeks, then 2/week for 36 weeks

Exclusion Criteria:

* History of any neurological, cardiovascular, or orthopedic condition that can limit their ability to participate
* Individuals who self-report engaging in more than 120 minutes of vigorous physical activity per week at baseline

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
. Functional Gait Assessment (FGA) | Assess the change between baseline and post 9-month intervention.
  FGA is a 10-item test, assessing walking and balance.It is well validated as a predictor for falls for people with PD

SECONDARY OUTCOMES:
6 minute walk test (6MWT)- | Assess the change between baseline and post 9-month intervention.
  6 MWT assesses physical endurance. Participants will be asked to walk down a hallway at a comfortable speed for 6 min.
Semi-structured interview | Assess the change between baseline and post 9-month intervention.
  To assess the attitude of participants toward the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Diana Krasteva, Bachelor's, Principal Investigator — Vancouver Coastal Health/ University of British Columbia
Locations (1):
- Lions Gate Hospital, North Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886